CLINICAL TRIAL: NCT00409253
Title: Treatment of Severe Hypertension During Pre-Eclampsia.A Preliminary Equivalence Study Between URAPIDIL and NICARDIPINE
Brief Title: Treatment of Severe Hypertension During Pre-Eclampsia: A Preliminary Equivalence Study Between Urapidil and Nicardipine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER, Direction de la Recherche Clinique et de l'Innovation - Hôpitaux Universitaires de Strasbourg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3738
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Hypertension During Pre-Eclampsia
Keywords: PRE-ECLAMPSIA-URAPIDIL-NICARDIPINE
MeSH Terms: interventions — urapidil; Nicardipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Urapidil (Active Comparator)
  Interventions: Drug: URAPIDIL (EUPRESSYL*)
- Nicardipine (Active Comparator)
  Interventions: Drug: NICARDIPINE

INTERVENTIONS:
Drug: URAPIDIL (EUPRESSYL*) — Urapidil (Eupressyl*) :IV (PSE) 1 microg/kg/min° until reduction PAM 15 %. Reduction ¼ of the posology to obtain PAM between 105 and 125 mmHg with adjustment 0.25 microg/kg/min/15 min. Maximal dose = 30mg/h.
  Arms: Urapidil
Drug: NICARDIPINE — Nicardipine : IV 6.25 mg bolus until PAD >105 mm/Hg. Perfusion (PSE) 4 mg/h to obtain PAM between 105 and 125 mm/Hg with adjustment 2mg/h/5 min without overshoot 20 mg/h Maximal treatment duration : 7 days
  Arms: Nicardipine

SUMMARY:
The aim of this study is to confirm that URAPIDIL is as efficient and as safe as NICARDIPINE to correct severe hypertension in pre-eclamptic patients.

* efficacy endpoint : mean arterial blood pressure corrected to 105-125 mmHg after 120 min of study drug administration.
* safety endpoints : clinical, biological and ultrasound observation for any side effect.All infants will be observed in the neonatology unit (during 48h).

ELIGIBILITY:
Inclusion criteria:

* patients 'written informed consent dated and signed by investigator and patient
* affiliation to a social security system
* single pregnancy
* arterial hypertension (PAS ≥140 and/or PAD≥90) in the context of severe pre-eclampsia

Exclusion criteria:

* patient under 18 year old or unable to give informed consent
* protocol rejected by patient-impossibility to use non invasive blood pressure monitoring
* antihypertensive treatments within 24h before inclusion
* allergy to or contraindication for one of the study drugs-pre
* eclampsia that does not require an antihypertensive treatment
* acute eclampsia-requirement for other drugs with potential dangerous interactions with study drugs
* participation to a therapeutic protocol within 6 months prior to the start of study

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Systolic, diastolic, mean blood pressure and pulse rate :-every 5 min during the titration phase-every 15 min up to the second hour treatment-every hour up to the 6th hour and every 3 hour during the rest of the treatment period. | Systolic, diastolic, mean blood pressure and pulse rate :-every 5 min during the titration phase-every 15 min up to the second hour treatment-every hour up to the 6th hour and every 3 hour during the rest of the treatment period

SECONDARY OUTCOMES:
-maternal and foetal ultrasonography, biology and clinical assessment-type of delivery-post-partum bleeding-neo-natal evaluation by neonatologist during the first 48 hours of life | During the first 48hour of life

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Auguste DIEMUNSCH, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (4):
- France (4):
  - Hôpital Saint-Jacques, CHU de Besançon, Besançon
  - Maternité A. PINARD, Nancy
  - Sihcus-Cmco, Schiltigheim
  - Service d'Anesthésie et de Réanimation Médicale, Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg

REFERENCES:
- [Derived] Diemunsch P, Garcia V, Lyons G, Pottecher J, Emmanuel S. Urapidil versus nicardipine in preeclamptic toxaemia: A randomised feasibility study. Eur J Anaesthesiol. 2015 Nov;32(11):822-3. doi: 10.1097/EJA.0000000000000303. No abstract available. PMID 26148170